CLINICAL TRIAL: NCT00594022
Title: The Effect of Vestibular Stimulation on Transient Insomnia Induced by a Five-hour Phase Advance of Sleep Time
Brief Title: Evaluation of Vestibular Stimulation to Help Occasional Sleeplessness
Acronym: VSOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MR-0707-VSOM-MS
Record Dates: First submitted 2007-12-26; First posted 2008-01-15 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Insomnia; Sleeplessness; Transient Insomnia
Keywords: Electric Stimulation; Latency to Persistent Sleep (LPS); Transient Insomnia; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1- "VirtuSom" - Stim (Active Comparator): Normal sleepers (7.5 - 9.0 hours), MSLT (multiple sleep latency test) >=14 min; phase-advance 5-hours studied under full polysomnogram (PSG) with active device (electric stimulation of the Vestibular nerve).
  Interventions: Device: Electric stimulation of the Vestibular Nerve - "VirtuSom"
- Group 2- "VirtuSom"- Sham (Placebo Comparator): Normal sleepers (7.5 - 9.0 hours), MSLT >=14 min; phase-advance 5-hours studied under full polysomnogram (PSG) with placebo / sham device (NO electric stimulation of the Vestibular nerve).
  Interventions: Device: Electric stim of the Vestibular Nerve - "VirtuSom" - SHAM

INTERVENTIONS:
Device: Electric stimulation of the Vestibular Nerve - "VirtuSom" — This device is similar to a Tens or Micro-Current electrical stimulator with respect to current levels deliver; however, because of the location of the stimulation it is similar to a Cranial Electrical Stimulator. A small electric stimulation (100 uA - 1000 uA) will be provided at the mastoids (bi-laterally) via small hydrogel electrodes.
  Arms: Group 1- "VirtuSom" - Stim
Device: Electric stim of the Vestibular Nerve - "VirtuSom" - SHAM — This device is similar to a Tens or Micro-Current electrical stimulator with respect to current levels deliver; however, because of the location of the stimulation it is similar to a Cranial Electrical Stimulator. For the Sham Group, NO electric stimulation (100 uA - 1000 uA) will be provided at the mastoids (bi-laterally) via small hydrogel electrodes. This is a sham / placebo device only.
  Arms: Group 2- "VirtuSom"- Sham

SUMMARY:
The purpose of this study is to determine whether a small electrical current to the vestibular nerve (balance organ) will decrease the time it take for participants to fall asleep.

DETAILED DESCRIPTION:
This 2 arm study will look at the proposed treatment (electrical stimulation of the vestibular nerve) versus a sham or placebo device. The effect of the device will be evaluated in a study that uses normal sleepers and advances them(puts them to bed 5-hours earlier than normal) to see if they fall asleep faster in one group or the other. Stimulation in the treated or sham group is only for the first hour after lights off.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 21- 50 attempts will be made to enroll equal distributions of males and females
* Able and willing to provide written informed consent
* Self reported habitual bedtime between 2100 and 0100 hours, which does not vary by more than 1 hour at least 5 nights per week
* Self reported 7.5-9 hrs. habitual sleep time
* Able to commit to 9 hrs of sleep opportunity throughout the study, but especially for the 3 nights prior to their PSG
* Pass Berlin questionnaire, i.e. low likelihood of sleep disordered breathing
* No history or evidence of RLS(restless leg syndrome) /PLMS (periodic limb movement syndrome) /Narcolepsy, no non-respiratory related sleep disorders.

Exclusion Criteria:

* Regular use of a pack or more per day of tobacco products
* Typically consumes more than 2 (12 oz) caffeinated beverages per day
* Self reported history of motion sickness
* Participation in a study of investigational or marketed drugs or devices during the 30-day period prior to the start of the study or during the study
* Clinically significant medical or psychiatric condition as determined by the investigator
* Probable diagnosis of a current sleep disorder including but not limited to insomnia, sleep apnea, restless legs syndrome, or periodic limb movement disorder
* History of current or recent (e.g. within past 5 years) alcohol, narcotic or any other drug abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, 4th Edition (DSM-IV)
* Currently works night shift or rotating shift
* Travel or planned travel across more than 1 time zone within one week prior to randomization
* Use of any medication that, in the opinion of the investigator, may alter sleep or wakefulness. (See Appendix E: Guideline For Medications Commonly Associated With Alterations Of Sleep / Wake Functioning). Subjects will undergo urine drug testing.
* Consumption of more than 14 alcoholic drinks per week, or the recent consumption of more than 4 alcoholic drinks in one night. Subjects will be tested for alcohol, using a saliva test kit.
* Pregnancy (will confirm absence of pregnancy with a urine or serum pregnancy test in women's of child bearing age).
* Presence of a pacemaker
* Presence of epilepsy or other uncontrolled medical conditions.
* Prior participation in a VirtuSom protocol
* History of vestibular disorders, (such as vertigo)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 349 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, Principal Investigator — Duke University Medical Center, Duke Clinic Sleep Lab
Locations (6):
- United States (6):
  - Neuro Trials, Atlanta, Georgia
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Clinilabs, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Tri-State Sleep Disorders Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1- "VirtuSom" - Stim: Normal sleepers (7.5 - 9.0 hours), MSLT >=14 min; phase-advance 5-hours studied under full polysomnogram (PSG) with active device (electric stimulation of the Vestibular nerve).
  Electric stimulation of the Vestibular Nerve - "VirtuSom": This device is similar to a Tens or Micro-Current electrical stimulator with respect to current levels deliver; however, because of the location of the stimulation it is similar to a Cranial Electrical Stimulator. A small electric stimulation (100 uA - 1000 uA) will be provided at the mastoids (bi-laterally) via small hydrogel electrodes.
Period: Overall Study
Arm/Group | Group 1- "VirtuSom" - Stim | Group 2- "VirtuSom"- Sham
Started | 176 | 173
Completed | 176 | 173
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1- "VirtuSom" - Stim | Group 2- "VirtuSom"- Sham | Total
Number analyzed (Participants) | 176 | 173 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.53 (7.56) | 31.91 (7.74) | 31.76 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 118 | 237
  Male | 57 | 55 | 112
Region of Enrollment [Number; unit: participants]
  United States | 176 | 173 | 349
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.42 (5.04) | 26.00 (5.42) | 25.71 (5.23)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 71.62 (8.86) | 72.84 (9.00) | 72.23 (8.94)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 113.57 (12.39) | 115.64 (11.91) | 114.60 (12.18)
Respiration [Mean (Standard Deviation); unit: breaths per minute] | 16.49 (2.19) | 16.82 (1.88) | 16.65 (2.05)
Pulse [Mean (Standard Deviation); unit: beats per minute] | 70.14 (9.99) | 69.43 (9.60) | 69.79 (9.79)
Sleep Onset Latency on Multiple Sleep Latency Test [Mean (Standard Deviation); unit: minutes] | 17.79 (1.90) | 17.93 (1.81) | 17.86 (1.86)

OUTCOME MEASURES:

1. Primary Outcome: Latency to Persistent Sleep (LPS)
Description: Latency to Persistent Sleep is how long does it take for a person to fall asleep and stay asleep. This is measured in minutes. This is different from sleep onset latency as participants fall asleep, but may wake back up.
Time Frame: Treatment Night
Population: Only 282 of the Polysomnography results were scorable. 132 for the treatment (stim group) and 150 for the sham group.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1- "VirtuSom" - Stim | Group 2- "VirtuSom"- Sham
Number analyzed (Participants) | 132 | 150
minutes | 48.14 (70.41) | 58.84 (87.03)
Statistical Analysis 1: Comparison: Group 1- "VirtuSom" - Stim vs Group 2- "VirtuSom"- Sham; Test type: Superiority or Other; p = .1275, t-test, 1 sided

2. Secondary Outcome: Subjective Sleep Onset Latency (SOL)
Description: Subjective sleep onset latency is how long it took a person to fall asleep once lights out. For subjective SOL this is a question to a participant the next morning asking how long they felt it took them to fall asleep in minutes.
Time Frame: Treatment night
Population: Site 6 indicate that there are properties of either the population or the study site that make it different from the remaining sites. For this reason, the analysis of the primary and secondary endpoints of the trial were done with Site 6 excluded.
  Not all participants answered this question the following morning, participants analyzed is less
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1- "VirtuSom" - Stim | Group 2- "VirtuSom"- Sham
Number analyzed (Participants) | 102 | 118
minutes | 79.16 (97.78) | 87.91 (101.16)

3. Secondary Outcome: Total Sleep Time (TST) in the First 2 Hours After Lights Out
Description: Total sleep time is the total amount of sleep a person gets in minutes over the course of the night. For this outcome measure it is for the 2 hours after lights out.
Time Frame: Treatment night
Population: It was noted on initial evaluation of the results, that Site 6 indicate that there are properties of either the population or the study site that make it different from the remaining sites. For this reason, the analysis of the primary and secondary endpoints of the trial were done with Site 6 excluded.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1- "VirtuSom" - Stim | Group 2- "VirtuSom"- Sham
Number analyzed (Participants) | 113 | 129
minutes | 66.65 (32.81) | 64.17 (36.75)

4. Secondary Outcome: Total Sleep Time (TST) in the First Hour After Lights Out
Description: Total sleep time is the total amount of sleep a person gets in minutes over the course of the night. For this outcome measure it is the total amount of sleep a participant gets over the first hour of sleep after lights out.
Time Frame: Treatment night
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1- "VirtuSom" - Stim | Group 2- "VirtuSom"- Sham
Number analyzed (Participants) | 113 | 129
minutes | 33.84 (16.01) | 30.51 (18.15)

5. Secondary Outcome: Scored Sleep Onset Latency (SOL on PSG)
Description: Sleep onset latency is the amount of time it takes to fall asleep after the lights have been turned off. For this outcome measure it is as measured by the scored PSG.
Time Frame: Treatment Night
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1- "VirtuSom" - Stim | Group 2- "VirtuSom"- Sham
Number analyzed (Participants) | 113 | 129
minutes | 27.50 (49.79) | 31.28 (50.03)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group 1- "VirtuSom" - Stim | Group 2- "VirtuSom"- Sham
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/173
Other Adverse Events (participants affected / at risk) | 9/176 | 11/173
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- "VirtuSom" - Stim (N=176) | Group 2- "VirtuSom"- Sham (N=173)
Headache (Nervous system disorders) | 9 (10) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No